CLINICAL TRIAL: NCT00147186
Title: The Effectiveness of Hylan GF-20 on Joint Reaction Forces and Kinematic Patterns During Gait in Patients With Knee Osteoarthritis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Kessler Foundation (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: 100653
Record Dates: First submitted 2005-09-06; First posted 2005-09-07 (Estimated); Last update posted 2007-01-15 (Estimated); Status verified 2005-06

CONDITIONS: Osteoarthritis
MeSH Terms: conditions — Osteoarthritis

INTERVENTIONS:
Device: Hylan G-F 20

SUMMARY:
The use of Hylan G-F 20 as a treatment of osteoarthritis (OA) of the knee has become popular in recent years. Typical treatment of OA of the knee includes NSAIDs and physical therapy protocols to strengthen local muscle groups and decrease pain. When these conservative treatment modalities have been exhausted, the next step is arthroplasty of the knee. Hylan G-F 20 treatments provide physicians with an intermediate mode of treatment prior to surgery. Hylan G-F 20 is a cross-linked, high molecular weight derivative of hyaluronan which can be found within the synovial capsule of the knee. This form of viscosupplementation is intended to reduce the pain suffered by those with OA by increasing the fluid levels within the synovial space, providing a cushion between the bony surfaces within the knee joint. Current studies have only looked at self-reported pain relief or Outcomes Inventories. This study aims to determine the ability of Hylan G-F 20 treatment to improve the parameters of gait of individuals who suffer from OA.

DETAILED DESCRIPTION:
Typically, when an adult suffers from OA of the knee, they are presented with two choices: conservative treatments consisting of NSAID therapy and physical therapy or surgical intervention to replace the affected knee joint. There is a third avenue of treatment that has become available in recent years. This treatment modality is viscosupplementation. Viscosupplementation consists of replacing hyaluronic acid in the synovial fluid contained in the knee joint. It has been observed that the synovial fluid of OA sufferers has less hyaluronic acid (HA), and the HA that remains is of lower molecular size and concentration Replacement of the HA contained in the synovial fluid through the use of Hylan G-F 20 has been shown in clinical studies to be clinically safe, and have the ability to provide pain relief with a minimum of adverse reactions. Clinical studies concerning the use of Hylan G-F 20 have focused on safety and efficacy in regards to pain relief in those who suffer OA. To date, there have been few studies performed looking at the efficacy of Hylan G-F 20 on the kinematics and kinetics of gait. This study will provide data on the ability of Hylan G-F 20 treatment to improve the temporal-spatial parameters of gait in those who suffer OA, as well as the ability of Hylan G-F 20 to reduce joint reaction forces in the affected knee.

ELIGIBILITY:
Inclusion Criteria:

* ambulatory, unilateral knee OA of at leas 3 months confirmed by radiography, pain requiring NSAIDS for at least 2 months

Exclusion Criteria:

* no trauma to target knee within last 5 years, prior viscosupplementation therapy, allergy to avian products, inflammatory disease, joint sepsis,varus/valgus >12 degrees, clinically apparent tense effusion, oral corticosteroids, intra-articular injection in any joint within the last 3 months, venous or lymphatic stasis in the leg, claudication or PVD, major surgery, arthroplasty in the target joint, arthroplasty in non-target knee within the last 6 months, current malignancy or treatment within the last 5 years, except for non-melanoma skin cancer, planned surgery during the study period, diabetes requiring insulin, use of an investigational device or drug (including glucosamine and chondroitin sulfate) within 90 days before entering the study, significant psychiatric or neurological disorder, active alcohol abuse or drug abuse within the past year.

Min Age: 41 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2000-01; Study Completion 2005-05

PRIMARY OUTCOMES:
Gait kinematics, kinetics, WOMAC, VAS

CONTACTS AND LOCATIONS:
Overall Officials: Sue A Sisto, Ph.D., PT, Principal Investigator — Kessler Medical Rehabilitation Research and Education Corporation
Locations (1):
- Kessler Medical Rehabilitation Research and Education Corporation, West Orange, New Jersey, United States